CLINICAL TRIAL: NCT05439525
Title: Effect of Mulligan on Sub-acromial Space in Patients With Shoulder Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.t.Rec/012/003613
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Shoulder Impingement
Keywords: mulligan technique; sub-acromial space
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: mulligan and conventional therapy
Who Masked: Outcomes Assessor
Masking Description: permuted block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): the patient will receive Shoulder complex mobilization with movement three time a week for two weeks
  Interventions: Other: mulligan technique; Other: conventional therapy
- Group B (Active Comparator): will receive Conventional therapy three times a week for two weeks.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: mulligan technique — The patient will be in sitting and the therapist stands on the contralateral side of pain, stabilizing the scapula posteriorly with one hand. The head of the humerus is translated posteriorly and laterally with the other hand, along the plane of the glenoid fossa. While the glide is sustained, the patient actively elevates their arm through the plane of abduction or scaption (elevation). Apply 6-10 repetitions in a set, with 3-5 sets in a treatment session the perform mobilization on acromioclavicular and sternoclavicular joint
  Arms: Group A
Other: conventional therapy — 1. Flexibility exercises: enhance flexibility of the glenohumeral Posterior capsule, pectoralis muscle, and upper thoracic spine.
  2. Strengthen the rotator cuff and scapular stabilizers.
  3. Improve upper-quarter postural awareness

SUMMARY:
the aim of this study is to investigate the Effect of mulligan technique on sub-acromial space in patients with shoulder impingement syndrome

DETAILED DESCRIPTION:
Shoulder Impingement Syndrome (SIS) is defined as the mechanical entrapment of the rotator cuff (mainly the supraspinatus tendon) or the sub-acromial bursa in the sub-acromial space between the humeral head and the acromion or coracohumeral ligament .It is typically exacerbate when the arm is elevated or when overhead throwing activities are performed . Mulligan technique is a type of manual therapy with hypoalgesic effects, increases joint ROM, enhances muscle function and treats specific pathologies. Mobilization with movement (MWM) can be defined as the application of a sustained passive accessory force / glide to a joint while the patient actively performs a task that was previously identified as being problem.

ELIGIBILITY:
Inclusion Criteria:

age of patients from 30- 55 years old . Both Male and female.

Shoulder pain and two out of four specified objective signs and symptoms:

Positive Neer impingement test. Positive Hawkins-Kennedy impingement test. Painful or limitation of active shoulder elevation (flexion, abduction, scaption).

Pain or limitation with the functional movement patterns of hand-behind-back or hand-behind-head.

Exclusion Criteria:

Systemic or neurological disorder. Adhesive capsulitis. Cervical radiculopathy. History of shoulder surgery. Corticosteroid injection within the past month Subjects who had received physical therapy treatment for their shoulder within the past three months.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-05 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
sub-acromial space | up to two weeks
  sub-acromial space will be measured by ultrasonography

SECONDARY OUTCOMES:
shoulder range of movement | up to two weeks
  shoulder range of motion will be measured by digital goniometer

OTHER OUTCOMES:
pressure pain threshold | up to two weeks
  pressure algometer will be used to measure pressure pain threshold
shoulder function | up to two weeks
  quick DASH will be used to measure shoulder function. DASH is a shortened version of the DASH questionnaire that uses 11 items to measure the degree of difficulty in performing various physical activities due to a shoulder, arm, or hand problem (6 items); the severity of pain and tingling (2 items); and the problem's effect on social activities, work, and sleep (3 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Cairo, Egypt